CLINICAL TRIAL: NCT01343472
Title: Evaluation of the Washington Intensive Supervision Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pepperdine University (Other)
Responsible Party: Principal Investigator, Brett T. Leach, Regulatory Affairs Specialist, Pepperdine University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPP0311F08
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Behavior; Drug Users
Keywords: Behavior; Drug users
MeSH Terms: conditions — Behavior; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WISP supervision (Experimental): Parolee supervised under WISP parole model.
  Interventions: Behavioral: WISP supervision
- Parole-as-usual (Active Comparator): Parolees supervised under Washington State's parole-as-usual
  Interventions: Behavioral: Parole-as-usual

INTERVENTIONS:
Behavioral: WISP supervision — WISP entails a warning session (Orientation Hearing) where the rules of parole are laid out and parolees are told that any violation of stated parole conditions will be sanctioned with a brief jail term (typically a few days in jail). WISP includes regular random drug testing.
  Other Names: HOPE supervision
  Arms: WISP supervision
Behavioral: Parole-as-usual — Parolees are supervised under standard parole supervision practice in Washington State.
  Other Names: PAU
  Arms: Parole-as-usual

SUMMARY:
This study entails an evaluation of the Washington Intensive Supervision Program (WISP). The purpose of the evaluation is to test whether subjects assigned to WISP perform better than those assigned to parole-as-usual (PAU).

DETAILED DESCRIPTION:
This study entails an evaluation of the Washington Intensive Supervision Program (WISP). WISP is a program targeting high-risk parolees in Seattle, and is modeled after the HOPE program in Hawaii. The purpose of the evaluation is to test whether subjects assigned to WISP perform better than those assigned to parole-as-usual (PAU) on a number of outcomes, including drug use, missed appointments, recidivism, prison and jail stays, and parole revocations. WISP uses regular random drug testing and close community supervision, paired with swift and certain, but modest sanctions for every detected violation.

ELIGIBILITY:
Inclusion Criteria:

* Inmates released by DOC to community corrections supervision
* Supervised out of the Seattle CJC (Community Justice Center) to include field offices and offenders from the downtown "Metro" unit, Southeast Seattle unit, Northgate (north Seattle) and West Seattle.
* Have a parole supervision discharge date at least one year from the date of release from entry into WISP

Exclusion Criteria:

* Level III Sex Offenders
* Existing assignment to supervision that precludes WISP. These include: Drug Offender Sentencing Alternative (DOSA)and Special Sex Offender Sentencing Alternative (SSOSA).
* Dangerously Mentally Ill (DMIO)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Revocation rate | 12 months
  Percentage of subjects in each condition who are revoked from parole and returned to prison

SECONDARY OUTCOMES:
% positive drug tests | 12 months
  Percentage of random and scheduled drug tests that test positive for illicit drugs
Days incarcerated | 12 months
  Total number of days incarcerated in jail or prison
% Missed appointments | 12 months
  Percentage of parole appointments that are missed.
New arrests | 12 months
  Number of new arrests.
Assessed risk | 12 months
  Parolee risk assessment (high, medium, low)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hawken, PHD, Principal Investigator — Pepperdine University
Locations (1):
- Seattle Community Justice Center, Seattle, Washington, United States